CLINICAL TRIAL: NCT04945018
Title: A Phase I/II Study of Human Induced Pluripotent Stem (iPS) Cell-derived Cardiomyocyte Spheroids (HS-001) in Patients With Severe Heart Failure, Secondary to Ischemic Heart Disease
Brief Title: A Study of iPS Cell-derived Cardiomyocyte Spheroids (HS-001) in Patients With Heart Failure (LAPiS Study)
Acronym: LAPiS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heartseed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-001-01
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Ischemic Heart Disease
Keywords: Heart Failure; Ischemic Heart Disease
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HS-001 Low dose (Experimental): HS-001 Low dose Administration
  Interventions: Biological: HS-001 CS; Device: HS-001-D needle, HS-001-D Adaptor
- HS-001 High dose (Experimental): HS-001 High dose Administration
  Interventions: Biological: HS-001 CS; Device: HS-001-D needle, HS-001-D Adaptor

INTERVENTIONS:
Biological: HS-001 CS — Human (allogeneic) iPS-cell-derived cardiomyocyte spheroids suspension
Device: HS-001-D needle, HS-001-D Adaptor — Cardiomyocyte spheroids Dedicated Needles for Implantation and Guided Adaptors

SUMMARY:
The purpose of this clinical study is to evaluate the safety and efficacy of HS-001 CS transplanted into severe heart failure patients with underlying ischemic heart disease for 26 weeks after transplantation.

DETAILED DESCRIPTION:
This is a multicenter, open-label, two-group dose-escalation, phase I/II study in 10 severe heart failure patients (five in the low-dose group and five in the high-dose group) with underlying ischemic heart disease.

After screening period is completed, subjects undergo HS-001 CS transplantation. After transplantation, subjects take immunosuppressant and have efficacy/safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resting left ventricular ejection fraction (LVEF) ≦40% based on institutional assessment on either screening cardiac MRI or echocardiographic assessment
* New York Heart Association (NYHA) cardiac function classification of grade II or higher at screening
* Other Criteria apply, please contact the investigator

Exclusion Criteria:

* Patients screened less than 1 month after the onset of myocardial infarction
* Patients with congenital heart disease, or cardiac sarcoidosis
* Other Criteria apply, please contact the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 26 weeks post-transplant
  Adverse events and safety in the 26 weeks after HS-001 CS transplantation

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction in Cardiac MRI scan & Echocardiography | 26 weeks and 52 weeks post-transplant
  Left Ventricular Ejection Fraction in the 26 weeks and 52 weeks after HS-001 CS transplantation
Myocardial wall motion evaluation in Echocardiography | 26 weeks and 52 weeks post-transplant
  Myocardial wall motion evaluation (Index of myocardial strain) in the 26 weeks and 52 weeks after HS-001 CS transplantation
Myocardial blood flow in SPECT | 26 weeks and 52 weeks post-transplant
  Myocardial blood flow in the 26 weeks and 52 weeks after HS-001 CS transplantation
Myocardial viability in SPECT | 26 weeks and 52 weeks post-transplant
  Myocardial viability in the 26 weeks and 52 weeks after HS-001 CS transplantation
6-minute walk distance | 26 weeks and 52 weeks post-transplant
  6-minute walk distance in the 26 weeks and 52 weeks after HS-001 CS transplantation
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 26 weeks and 52 weeks post-transplant
  Kansas City Cardiomyopathy Questionnaire in the 26 weeks and 52 weeks after HS-001 CS transplantation
5-level EQ-5D version (EQ-5D-5L) | 26 weeks and 52 weeks post-transplant
  5-level EQ-5D version (EQ-5D-5L) in the 26 weeks and 52 weeks after HS-001 CS transplantation
N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) | 26 weeks and 52 weeks post-transplant
  N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) in the 26 weeks and 52 weeks after HS-001 CS transplantation

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - St. Marianna University Hospital, Kawasaki
  - Saitama Medical University International Medical Center, Saitama
  - Juntendo University Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Tokyo Medical and Dental University Medical Hospital, Tokyo
  - Tokyo Metropolitan Geriatric Medical Center, Tokyo
  - Tokyo Women's Medical University, Tokyo

IPD SHARING:
Plan to Share IPD: No